CLINICAL TRIAL: NCT01453322
Title: Video Documentation of Localized Complications in IV Cannulation Using Near-Infrared Technology
Brief Title: Video Documentation of Localized Complications
Status: Completed | Type: Observational
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP1009
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Vascular Access
Keywords: Veins; Vascular Access; IV complications; VeinViewer Vision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to confirm and document that with the use of a FDA Class I exempt near infrared device, VeinViewer® Vision that is hands-free and can be used for healthy adult volunteers with varying skin types to assist in the improved visualization, it is possible to film, analyze and document PIV localized complications and venous flow and refill.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be considered in good health by investigator
* Must be able to read and understand English

Exclusion Criteria

* Less than 18 years of age
* Known allergy to Heparin
* History of HIT (Heparin-induced thrombocytopenia)
* Unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Valve and Refill Confirmation | Immediately after flush-Day 1
  Using VeinViewer, the clinician will be able to view valves and refill. It will be confirmed using Ultrasound.

SECONDARY OUTCOMES:
Video Documentation of localized vascular access complications | Immediately after attempt-Day 1
  Using VeinViewer, the user will be able to detect hematomas and infiltrations.

CONTACTS AND LOCATIONS:
Overall Officials: Edward P Scott, MD, Principal Investigator — Key Biologics, LLC
Locations (1):
- Key Biologics LLC, Memphis, Tennessee, United States